CLINICAL TRIAL: NCT00223977
Title: A Multi-center, Randomized, Open Label Study of the Efficacy and Safety of Two Doses of Ferrlecit Versus Oral Iron to Treat Iron-deficiency Anemia in Peroneal Dialysis Patients Receiving Erythropoietin.
Brief Title: 2 Doses of Ferrlecit Versus Oral Iron to Treat Iron-deficiency Anemia in Peritoneal Dialysis Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR03001
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Anemia.
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferric gluconate; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sodium ferric gluconate complex 125 mg (Experimental): 125 mg sodium ferric gluconate weekly x 8 weeks
  Interventions: Drug: Sodium Ferric Gluconate Complex
- Sodium ferric gluconate complex 250 mg (Experimental): 250 mg sodium ferric gluconate complex weekly x 4 weeks
  Interventions: Drug: Sodium Ferric Gluconate Complex
- Oral iron (Active Comparator): 325 mg ferrous sulfate three times daily x 8 weeks
  Interventions: Drug: Oral Iron

INTERVENTIONS:
Drug: Sodium Ferric Gluconate Complex — 125 mg weekly x 8 weeks
  Other Names: Ferrlecit
  Arms: Sodium ferric gluconate complex 125 mg
Drug: Sodium Ferric Gluconate Complex — 250 mg weekly x 4
  Other Names: Ferrlecit
  Arms: Sodium ferric gluconate complex 250 mg
Drug: Oral Iron — 325 mg ferrous sulfate orally three times daily x 8 weeks
  Arms: Oral iron

SUMMARY:
This is a phase 3 clinical investigation. Patients who meet the eligibility criteria and provide signed informed consent will be randomized to receive one of two levels of Ferrlecit or oral iron in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Received maintenance peritoneal dialysis therapy for at least 4 weeks.
* Was expected to remain on peritoneal dialysis therapy for duration of study.
* Had predetermined low hemoglobin and transferrin saturation (TSAT) levels.
* Signed patient informed consent.

Exclusion Criteria:

* Had a predetermined serum levels of Ferritin and TSAT
* Pregnant or lactating.
* Had a serious concomitant medical disorder incompatible with participation in the study.
* Had a known hypersensitivity to Ferrlecit or any of its components.
* Unable to cooperate or comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2003-12; Primary Completion 2004-11 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hoel, RPh, PhD, Study Chair — Watson Pharmaceuticals
Locations (43):
- United States (19):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Los Angeles, California
  - Torrance, California
  - New Haven, Connecticut
  - Evanston, Illinois
  - Shreveport, Louisiana
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Royal Oak, Michigan
  - St Louis, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Sioux Falls, South Dakota
  - Dallas, Texas
  - Richmond, Virginia
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (5):
  - Kelowna
  - Kitchener
  - London
  - Scarborough
  - Toronto
- Zagreb, Croatia
- India (7):
  - Bangalore
  - Chandigarh
  - Chennai
  - Hyderabad
  - Lucknow
  - Mahīm
  - New Delhi
- Mexico (6):
  - Col. Toriello Guerra
  - Durango
  - Mexico City
  - Monterrey
  - Tlalpan
  - Zapopan
- Osijek, Poland
- Russia (2):
  - Moscow
  - Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Started | 46 | 58 | 42
Completed | 37 | 47 | 39
Not Completed | 9 | 11 | 3
Not completed — Adverse Event | 7 | 10 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron | Total
Number analyzed (Participants) | 46 | 58 | 42 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 53 | 35 | 122
  >=65 years | 12 | 5 | 7 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (14.11) | 48.1 (12.49) | 51.5 (12.88) | 50.5 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 27 | 80
  Male | 23 | 28 | 15 | 66
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 10
  Mexico | 6 | 8 | 9 | 23
  Poland | 8 | 9 | 7 | 24
  Croatia | 4 | 8 | 4 | 16
  Bulgaria | 1 | 3 | 1 | 5
  Russian Federation | 19 | 19 | 14 | 52
  India | 5 | 7 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin
Description: Change from baseline to 1 week after the last oral iron dose or 2 weeks after the last sodium ferric gluconate injection
Time Frame: Baseline to 5 weeks and 9 weeks
Population: modified intent to treat (mITT) with last observation carried forward (LOCF) imputation
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Number analyzed (Participants) | 46 | 55 | 42
ng/mL | 1.49 (1.09) | 0.89 (1.35) | 1.02 (1.55)

2. Secondary Outcome: Change From Baseline in Hematocrit (Hct)
Description: as for outcome 1
Time Frame: Baseline to 5 weeks and 9 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Number analyzed (Participants) | 46 | 55 | 42
percent | 4.62 (3.37) | 2.93 (4.61) | 3.07 (4.59)

3. Secondary Outcome: Change From Baseline in Transferrin Saturation (TSAT).
Description: as for outcome 1
Time Frame: Baseline to 5 weeks and 9 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Number analyzed (Participants) | 46 | 55 | 42
percent | 8.13 (8.77) | 8.2 (9.31) | 1.84 (6.5)

4. Secondary Outcome: Change From Baseline in Serum Ferritin.
Description: as for outcome 1
Time Frame: Baseline to 5 weeks and 9 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Number analyzed (Participants) | 46 | 55 | 42
ng/mL | 259.88 (212.73) | 368.67 (270.05) | 26.98 (86.57)

5. Secondary Outcome: Responders by Treatment Group
Description: Patients were classified as responders to treatment if they had an increase in Hgb of at least 1.0 g/dL assessed at 2 weeks following the final administration of Ferrlecit or 1 week following the last dose of oral iron.
Time Frame: Baseline to 5 weeks and 9 weeks
Measure: Number; unit: participants
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Number analyzed (Participants) | 46 | 55 | 42
participants | 30 | 22 | 20

ADVERSE EVENTS:
Arm/Group | Sodium Ferric Gluconate Complex 125 mg | Sodium Ferric Gluconate Complex 250 mg | Oral Iron
Serious Adverse Events (participants affected / at risk) | 3/46 | 13/58 | 7/42
Other Adverse Events (participants affected / at risk) | 16/46 | 20/58 | 12/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Ferric Gluconate Complex 125 mg (N=46) | Sodium Ferric Gluconate Complex 250 mg (N=58) | Oral Iron (N=42)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
CELLULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASC ACCID (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
EDEMA LUNG (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
FEVER (General disorders) | 0 (0) | 0 (0) | 1 (1)
FIBRILLAT ATR (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
HEM RECTAL (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCEM (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
HYPERVOLEM (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENS (Cardiac disorders) | 0 (0) | 5 (5) | 0 (0)
INFARCT MYOCARD (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
INJECT SITE REACT (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
KETOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (General disorders) | 2 (2) | 5 (5) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ULCER STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMIT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Ferric Gluconate Complex 125 mg (N=46) | Sodium Ferric Gluconate Complex 250 mg (N=58) | Oral Iron (N=42)
LAB TEST ABNORM (Blood and lymphatic system disorders) | 9 (11) | 8 (8) | 2 (2)
HYPERTENS (Cardiac disorders) | 4 (4) | 6 (6) | 4 (4)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (4)
HYPOTENS (Cardiac disorders) | 1 (2) | 4 (6) | 0 (0)
INFECT (General disorders) | 2 (2) | 1 (1) | 3 (3)
PAIN ABDO (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
PAIN (General disorders) | 0 (0) | 3 (4) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Primary endpoint for the 250 mg dose was 4 weeks earlier than the endpoint for the 125 mg dose, which may have contributed to lower Hbg increase with the 250 mg dose at endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less